CLINICAL TRIAL: NCT04884633
Title: Novel Method of Pancreatic Islet Transplantation Into the Omentum
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Frantisek Saudek (Other Government)
Responsible Party: Sponsor-Investigator, Frantisek Saudek, MD., prof., Institute for Clinical and Experimental Medicine
Organization: Institute for Clinical and Experimental Medicine (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-29009A
Record Dates: First submitted 2021-04-22; First posted 2021-05-13 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Islets of Langerhans Transplantation
Keywords: Pancreatic islets; Transplantation; Diabetes; Omentum
MeSH Terms: conditions — Diabetes Mellitus | interventions — Islets of Langerhans Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Pancreatic islet transplantation — New method of pancreatic islet transplantation into the omentum using a biodegradable scaffold

SUMMARY:
The investigators propose to conduct a pilot clinical study in 10 type 1 diabetic subjects suffering from hypoglycemia unawareness syndrome and episodes of severe hypoglycemia, in which therapy with transplantation of allogeneic pancreatic islets would be indicated according to current criteria at the Institute for Clinical and Experimental Medicine (IKEM). Pancreatic islets will be isolated and prepared for transplantation using the established laboratory technique with minor modifications corresponding to latest knowledge. In contrast to present routine, the islet preparation will not be administered percutaneously into the portal vein but will be placed on the surface of an omental pouch using a (mini) laparoscopic approach. Cell adherence will be achieved by addition of clinical-grade human thrombin that reacts with plasma to create a biocompatible, degradable gel containing the islet graft. The study will be performed in close collaboration with the Diabetes Research Institute (DRI) in Miami, which will provide expert assistance and technical training if needed.

DETAILED DESCRIPTION:
Despite continuing progress in pharmacological insulin substitution, insulin administration and monitoring of glucose levels, type 1 diabetes has been still associated with specific late organ complications. While the main pathophysiological factor for their development is chronic hyperglycemia, the critical limiting factor for achieving normal or near-normal blood glucose levels remains to be the risk of hypoglycemia. Stable glucose levels near the normal range maintained without the fear of low excursions have been so far achieved only by organ pancreas or islet transplantation, however at the cost of surgical procedure and lifelong immunosuppression to prevent rejection of the graft and recurrence of the autoimmune process. Transplantation is therefore considered only in patients with serious complications of diabetes in whom the quality of life is unacceptable. This group now includes also subjects with hypoglycemia unawareness syndrome complicated by severe life-threatening hypoglycemic episodes, in whom qualified medical treatment including available technological support failed.

Most islet transplantations are currently performed by a minimally invasive technique via infusion into the portal vein with subsequent seeding in the liver. This way of implantation, however, still bares significant risks of bleeding during the percutaneous portal catheterization or portal thrombosis. Several other factors suggest that the liver may not be the optimal site for islet infusion.

The optimal place for the islet graft should be based on minimally-invasive transplant procedure, allow to use relatively large volumes of tissue (e.g., for low purity preparations), enable noninvasive longitudinal monitoring and access for biopsy. Portal blood drainage would be preferable to reproduce physiological metabolic responses.

These requirements might fulfill implantation into the omentum as it represents a large, well-vascularized surface and the capillary beds lie directly under the mesothelium. Omentum is easily accessible and venous blood is drained into the portal system (as from the native islets). A technique for human islet transplantation into the omentum has recently been developed in the Diabetes Research Institute in Miami under the leadership of C. Ricordi. The Miami group demonstrated, that the islets re-suspended in either donor or autologous plasma and distributed in the omental pouch did not stick together and allowed regular distribution on the omentum surface. Better cell adherence was achieved by addition of clinical-grade human thrombin which supported development of a biocompatible, degradable gel containing the islet graft. This technology, which does not include any ex vivo biological manipulation with the islet cells (and does not therefore fall under the term "modern therapy" in EU], does not require the use of any officially yet not approved drugs or medical instruments, could be directly applied in a pilot clinical experiment and help to speed up the development of a more efficient and safer method for islet transplantation in type 1 diabetic subjects.

The investigators propose to conduct a pilot clinical study in 10 type 1 diabetic subjects suffering from hypoglycemia unawareness syndrome and episodes of severe hypoglycemia, in which therapy with transplantation of allogeneic pancreatic islets would be indicated according to current criteria at the Institute for Clinical and Experimental Medicine (IKEM). Pancreatic islets will be isolated and prepared for transplantation using the established labora¬tory technique with minor modifications corresponding to latest knowledge. In contrast to present routine, the islet preparation will not be administered percutaneously into the portal vein but will be placed on the surface of an omental pouch using a (mini) laparoscopic approach. Cell adherence will be achieved by addition of clinical-grade human thrombin that reacts with plasma to create a biocompatible, degradable gel containing the islet graft. Study procedures will be based on the protocol developed by the DRI with modifications resulting from experience of the applicant´s team and equipment of local facilities.

It is expected to include altogether 10 type-1 diabetic subjects with either

1. problematic hypoglycemia refractory to medical therapy including intensive insulin therapy, education and use of technological aids, or 2. end-stage kidney disease, who are eligible for kidney transplantation, but not eligible for whole organ pancreas transplantation due to a too high surgical risk

Inclusion criteria (in brief) The inclusion and exclusion criteria of the study meet the standard inclusion and exclusion criteria for islet transplantation with the following specifications and are listed (abbreviated) in the Eligibility section. Excluded will be subjects with Body Mass Index (BMI) >30 kg/m2 or patient weight ≤50 kg and glomerular filtration rate <80 mL/min/1.73 m2. Additional exclusion criteria specified in the full protocol.

Islet isolation from a compatible donor will be performed following standardized isolation protocol used in IKEM. The islets will be cultivated for up to 36 hours at 37°C in CMRL medium without any biological modification. The eligibility of the candidate will be reassessed by clinical and laboratory examination. Should a sufficient amount of islets (allowing to transplant 4000 IEQ/kg of the recipient) be obtained, the candidate will be prepared for the surgical mini-laparotomy procedure and the induction immunosuppressive therapy will be initiated.

After cultivation the islet cells will be collected, centrifuged, and after removing the su-pernatant, reconstituted in recipient's own plasma, the final ratio being 2:1 plasma to pellet. The operation will be conducted in general anesthesia by laparoscopic approach or under general anesthesia during the kidney transplant procedure (combined islet and kidney transplantation). The islet suspension will be aspired with a pipette and distributed on a suitable part of the omental surface (approx. 9x9 cm). Human thrombin, reconstituted from routinely used "surgical glue" preparation Tisseel Lyo® (Baxter) (or by another clinically approved preparation of thrombin) approximately in the same volume as the islet suspension, will be spread as another layer onto the islets to promote formation of a biodegradable gel containing the islet graft. This should facilitate the adherence to the omental surface and prevent the islets of pelleting. Omentum will then be gently folded to create a pouch and secured in place with stiches if necessary. The operation should last no more than 1-2 hours. The patients will be followed at the intensive care unit for a short time after the surgery with subsequent care at the intermediate care unit as usual after islet transplantation.

As for the immunosuppression regimen, the induction will consist of 3 doses of anti-T-lymphocyte globulin starting the day before transplant. Prophylactic immunosuppression will consist of a combination of tacrolimus (target trough levels 10-12 ng/ml tapered after 3 months to 6-10 ng/ml) and mycophenolate mofetil (1-2 g per day). In addition, etanercept (a TNF-α inhibitor) will be administered before the transplant (50 mg sc.) with subsequent doses of 25 mg on day 3, 7 and 10. Only a single dose of corticosteroids will be used before the first ATG infusion. All these drugs represent standard medical therapy after pancreas or islet transplantation in IKEM. A standard antibiotic and antiviral therapy will be administered according to the local policy in IKEM.

Blood glucose will be closely monitored and insulin administered with the aim to achieve near-normal glucose levels to prevent islet exhaustion. Continuous subcutaneous glucose monitors will be used after the dismissal from the hospital.

The post-transplant study follow-up will include 16 clinical visits. In addition, the recipients will be medically supervised as needed.

The clinical trial will aim at testing the safety and efficacy of the transplantation method. The primary safety endpoint will be demonstrating patient ´s safety throughout all stages of the trial. Primary efficacy endpoints will be achieving glycosylated HbA1c 53 mmol/mol at 1 year post-transplant and no severe hypoglycemia events from day 28 to 365 inclusive after the islet transplant.

Secondary efficacy endpoints (in brief) will be the following: the percent of reduction in insulin requirement, HbA1c levels, and response of C-peptide to stimulation by mixed meal test. Glucose variability and hypoglycemia duration data acquired from the continuous glucose monitoring system, quality of life measures (SF 36 questionnaire and diabetes treatment satisfaction questionnaire). Standard procedures to evaluate the quality of diabetes control (HYPO score, Clarke score, mixed meal test).

Secondary safety endpoints: Safety, including incidence of post-transplant infections, malignancies, morbidity, and other AEs (e.g., increased body weight and hypertension) associated with conventional immunosuppression. Renal function as measured by serum creatinine, GFR and other relevant laboratory parameters. Lipid profiles (triglycerides, total cholesterol, LDL cholesterol, HDL cholesterol) over time.

Assessment of the incidence and severity of adverse effects related to the transplantation procedure and immunosuppressive therapy.

Statistical evaluation Insulin needs will be estimated from the one-week self-report values. Estimates of population means and confidence intervals for those means will be reported for each follow-up visit. Numbers of severe hypoglycemic events will be estimated from the self-report values obtained at each follow-up visit. HbA1c and serum creatinine levels will be measured at study entry and at each follow-up visit. GFR will be estimated using the updated CKD-MDRD method. Estimates of population means and confidence intervals for those means will be reported for each follow-up visit. Linear mixed model methods will be used to describe trends with time. Incidence of serious adverse experiences will be tabulated by body system and graded by international Terminology Criteria for Adverse Events. In animal experiments islet survival rates (fed normoglycemia), areas under the curves of blood glucose and insulin during the intraperitoneal glucose tolerance test will be compared between the groups using nonparametric Wilcoxon and Mann-Whithey tests and Caplan-Mayer survival plots if applicable.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 to 65 years, ability to comply with the procedures of the study protocol.
* Clinical history of type 1 diabetes with onset at < 40 years of age, insulin-dependence for > 5 years at the time of enrollment.
* Absent stimulated C-peptide (<0,3 ng/l) in response to mixed meal test measured at 60 and 90 minutes after the start of consumption.
* Involvement in intensive diabetes management, defined as self-monitoring of glucose values no less that mean of three times each day averaged over each week and by the administration of three or more insulin injections each day or in-sulin pump. Management under the direction of a diabetologist with at least 3 clin¬ical evaluations during the12 months prior to study enrollment.
* At least on episode of severe hypoglycemia in the 12 months prior to the study enrollment
* Reduced awareness of hypo glycaemia (as specified in detail in the full protocol) during the screening period OR marked glycemic lability characterized by wide swings in blood glucose despite optimal diabetes therapy

Exclusion Criteria:

* Body Mass Index (BMI) >30 kg/m2 or patient weight ≤50 kg.
* Insulin requirement of >1.0 IU/kg/day or <15 U/day.
* glomerular filtration rate <80 mL/min/1.73 m2
* Additional exclusion criteria specified in the full protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2019-08-15 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 1 year
  The rate of serious adverse events
Achieving good metabolic control of diabetes | 1 year
  achieving glycosylated HbA1c 53 mmol/mol at 1 year post-transplant and no severe hypoglycemia events from day 28 to 365 inclusive after the islet transplant.

SECONDARY OUTCOMES:
Insulin requirement | 6 and 12 months
  The number of recipients with reduction of insulin dose by 50 percent or more
C-peptide | 6 and 12 months
  The number of recipients with C-peptide response to stimulation by mixed meal test over 0.5 pmol/ml
Quality of life assessed by the Short Form 36 questionnaire score | 12 months
  Evaluation of the Quality of Life Questionnaire SF 36 and comparison the score with th pre-transplant status (only observational outcome) Diabetes treatment satisfaction questionnaire
Infections | 1 year
  The number of recipients with severe or moderate treatment-related infections
The rate of significat glomerula filtration rate reduction | 6 months and 1 year
  The number of recipients with a reduction of the estimated glomerular filtration rate (eGFR) by 30 percent or more as compared with the pretransplant level

CONTACTS AND LOCATIONS:
Overall Officials: Frantisek Saudek, Principal Investigator — Institute for Clinical and Experimental Medicine
Locations (1):
- Institute for Clinical and Experimental Medicine, Department of Diabetes, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No